CLINICAL TRIAL: NCT01666314
Title: A Study in Japan and Ex-Japan to Characterize the Pharmacokinetic and Pharmacodynamic Response to Orteronel (TAK-700) in Chemotherapy-Naive Patients With Castration-Resistant Prostate Cancer
Brief Title: Study in Japan and Ex-Japan to Characterize the Pharmacokinetic and Pharmacodynamic Response to Orteronel (TAK-700) in Chemotherapy-Naive Participants With Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C21013; 2012-001539-30 (EudraCT Number); U1111-1179-5750 (Other: WHO)
Record Dates: First submitted 2012-08-06; First posted 2012-08-16 (Estimated); Results first posted 2018-03-20 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-02

CONDITIONS: Prostate Cancer
Keywords: castrate resistant prostate cancer,; CRPC,; orteronel,; TAK-700
MeSH Terms: conditions — Prostatic Neoplasms | interventions — orteronel; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Placebo + Orteronel 200 mg (Japan) (Other): Orteronel placebo-matching tablets, orally, twice daily in Cycle 1 (28 days) followed by orteronel 200 mg, tablets, orally, twice daily in 28 day cycles in Japan for up to 3.1 years. Study drug will be administered concomitantly with prednisone (or commercially available equivalent) 5 mg twice daily (BID) continuously throughout the study.
  Interventions: Drug: Orteronel; Drug: Orteronel Placebo; Drug: Prednisone
- Orteronel 200 mg (Japan) (Experimental): Orteronel 200 mg, tablets, orally, twice daily in 28 day cycles in Japan for up to 3 years. Study drug will be administered concomitantly with prednisone (or commercially available equivalent) 5 mg twice daily (BID) continuously throughout the study.
  Interventions: Drug: Orteronel; Drug: Prednisone
- Placebo + Orteronel 300 mg (Japan) (Other): Orteronel placebo-matching tablets, orally, twice daily in Cycle 1 followed by orteronel 300 mg, tablets, orally, twice daily in 28 day cycles in Japan for up to 2.8 years. Study drug will be administered concomitantly with prednisone (or commercially available equivalent) 5 mg twice daily (BID) continuously throughout the study.
  Interventions: Drug: Orteronel; Drug: Orteronel Placebo; Drug: Prednisone
- Orteronel 300 mg (Japan) (Experimental): Orteronel 300 mg, tablets, orally, twice daily in 28 day cycles in Japan for up to 2.8 years. Study drug will be administered concomitantly with prednisone (or commercially available equivalent) 5 mg twice daily (BID) continuously throughout the study.
  Interventions: Drug: Orteronel; Drug: Prednisone
- Placebo + Orteronel 200 mg (Ex-Japan) (Other): Orteronel placebo-matching tablets, orally, twice daily in Cycle 1 followed by orteronel 200 mg, tablets, orally, twice daily in 28 day cycles outside of Japan (Ex-Japan) for up to 3.1 years.
  Study drug will be administered concomitantly with prednisone (or commercially available equivalent) 5 mg twice daily (BID) continuously throughout the study.
  Interventions: Drug: Orteronel
- Orteronel 200 mg (Ex-Japan) (Experimental): Orteronel 200 mg, tablets, orally, twice daily in 28 day cycles Ex-Japan for up to 3.1 years. Study drug will be administered concomitantly with prednisone (or commercially available equivalent) 5 mg twice daily (BID) continuously throughout the study.
  Interventions: Drug: Orteronel; Drug: Prednisone
- Placebo + Orteronel 400 mg (Ex-Japan) (Other): Orteronel placebo-matching tablets, orally, twice daily in Cycle 1 followed by orteronel 400 mg, tablets, orally, twice daily in 28 day cycles Ex-Japan for up to 3.1 years. Study drug will be administered concomitantly with prednisone (or commercially available equivalent) 5 mg twice daily (BID) continuously throughout the study.
  Interventions: Drug: Orteronel; Drug: Orteronel Placebo; Drug: Prednisone
- Orteronel 400 mg (Ex-Japan) (Experimental): Orteronel 400 mg, tablets, orally, twice daily in 28 day cycles Ex-Japan for up to 3.1 years. Study drug will be administered concomitantly with prednisone (or commercially available equivalent) 5 mg twice daily (BID) continuously throughout the study.
  Interventions: Drug: Orteronel; Drug: Prednisone

INTERVENTIONS:
Drug: Orteronel — Orteronel tablets
Drug: Orteronel Placebo — Orteronel placebo-matching tablets
  Arms: Placebo + Orteronel 200 mg (Japan); Placebo + Orteronel 300 mg (Japan); Placebo + Orteronel 400 mg (Ex-Japan)
Drug: Prednisone — Prednisone 5 mg
  Arms: Orteronel 200 mg (Ex-Japan); Orteronel 200 mg (Japan); Orteronel 300 mg (Japan); Orteronel 400 mg (Ex-Japan); Placebo + Orteronel 200 mg (Japan); Placebo + Orteronel 300 mg (Japan); Placebo + Orteronel 400 mg (Ex-Japan)

SUMMARY:
This is a double-blind, placebo-controlled, multiregional Phase1/2 study to characterize the pharmacokinetic and pharmacodynamic responses to orteronel when administered concomitantly with prednisone in Chemotherapy-Naive Participants With Castration-Resistant Prostate Cancer

DETAILED DESCRIPTION:
The drug being tested in this study is called orteronel. Orteronel is being tested to treat adult males who have adenocarcinoma of the prostate. This study will look at the pharmacokinetics (how the drug moves through the body) and pharmacodynamics (how the drug effects the body) in people who take orteronel in addition to prednisone.

The study will enroll approximately 144 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the eight treatment groups (4 in Japan, 4 in Ex-Japan) which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need).

In Japan:

Participants were randomized in a ratio of 2:1:2:1

* 200 mg orteronel or Placebo-matching orteronel [(dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient] twice daily (BID) + prednisone
* 300 mg orteronel, or Placebo-matching orteronel, BID + prednisone Ex-Japan Participants were randomized in a ratio of 2:1:2:1
* 200 mg orteronel or Placebo-matching orteronel, BID in Cycle 1 + prednisone
* 400 mg orteronel, or Placebo-matching orteronel ,BID in Cycle 1 + Prednisone

Participants initially randomized to placebo received 4 weeks of placebo and then 12 weeks of active treatment with orteronel then entered a follow-up period treatment period. Participants initially randomized to orteronel received 16 weeks of treatment then entered a follow-up treatment period.

This multi-centre trial will be conducted worldwide. The overall time to participate in this study is approximately 3.2 years. Participants will make multiple visits to the clinic and a final visit 30 to 40 days after receiving their last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Male participants 18 years or older
* Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care
* Histologically or cytologically confirmed diagnosis of prostate adenocarcinoma
* Prior surgical castration or concurrent use of an agent for medical castration [e.g. Gonadotropin-releasing hormone (GnRH) analogue]
* Prostate-Specific Antigen (PSA) ≥ 2 ng/mL at screening
* Progressive disease based on PSA and/or radiographic criteria

Exclusion Criteria:

* Prior therapy with orteronel, ketoconazole, aminoglutethimide, or abiraterone.
* Known hypersensitivity to compounds related to orteronel, orteronel excipients, prednisone (or commercially available equivalent), or GnRH analogue.
* All antiandrogen therapy (including bicalutamide) is excluded within 4 weeks before the first dose of study drug. Any other therapies for prostate cancer, other than GnRH analogue therapy, such as progesterone, medroxyprogesterone, progestins (megesterol), or 5- alpha reductase inhibitors (e.g., finasteride or dutasteride), must be discontinued 2 weeks before the first dose of study drug.
* Continuous daily use of oral prednisone (or commercially available equivalent), oral dexamethasone, or other systemic corticosteroids for more than 2 weeks within the 3 months before screening (inhaled, nasal, and local steroids [e.g., joint injection] are allowed).
* Prior chemotherapy for prostate cancer, with the exception of neoadjuvant/adjuvant therapy as part of initial primary treatment for local disease that was completed 2 or more years before screening.

Please note that there are additional inclusion and exclusion criteria. The study center will determine if you meet all of the criteria.

Site personnel will explain the trial in detail and answer any question you may have if you do qualify for the study. You can then decide whether or not you wish to participate. If you do not qualify for the trial, site personnel will explain the reasons.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2012-08-20 (Actual); Primary Completion 2013-09-12 (Actual); Study Completion 2016-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- Urology Cancer Center, PC, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 43 investigative sites in Japan, United States, Greece, Australia, Netherlands, Ireland and United Kingdom from 20 August 2012 to 01 September 2016.
Pre-assignment Details: Male participants with a diagnosis of adenocarcinoma of the prostate were enrolled in the study. In Japan, participants were randomized to 200 mg orteronel, Placebo, 300 mg orteronel, or Placebo, BID, in a ratio of 2:1:2:1; ex-Japan participants were randomized to 200 mg orteronel, Placebo, 400 mg orteronel, or Placebo, BID, in a ratio of 2:1:2:1.
Groups:
- Placebo + Orteronel 200 mg (Japan): Orteronel placebo-matching tablets or Orteronel 200 mg, tablets, orally, twice daily (BID) in Cycle 1 (28 days) followed by orteronel 200 mg, tablets, orally, twice daily in 28 day cycles in Japan for up to 3 years. Study drug will be administered concomitantly with prednisone (or commercially available equivalent) 5 mg twice daily continuously throughout the study.
- Placebo + Orteronel 300 mg (Japan): Orteronel placebo-matching tablets or Orteronel 300 mg, tablets, orally, twice daily in Cycle 1 followed by orteronel 300 mg, tablets, orally, twice daily in 28 day cycles in Japan for up to 2.8 years. Study drug will be administered concomitantly with prednisone (or commercially available equivalent) 5 mg twice daily (BID) continuously throughout the study.
- Placebo + Orteronel 200 mg (Ex-Japan): Orteronel placebo-matching tablets, or Orteronel 200 mg, tablets, orally, twice daily in Cycle 1 followed by orteronel 200 mg, tablets, orally, twice daily in 28 day cycles outside of Japan (Ex-Japan) for up to 3.1 years. Study drug will be administered concomitantly with prednisone (or commercially available equivalent) 5 mg twice daily (BID) continuously throughout the study.
- Placebo + Orteronel 400 mg (Ex-Japan): Orteronel placebo-matching tablets, or Orteronel 400 mg, tablets, orally, twice daily in Cycle 1 followed by orteronel 400 mg, tablets, orally, twice daily in 28 day cycles Ex-Japan for up to 3.1 years. Study drug will be administered concomitantly with prednisone (or commercially available equivalent) 5 mg twice daily (BID) continuously throughout the study.
Period: Overall Study
Arm/Group | Placebo + Orteronel 200 mg (Japan) | Placebo + Orteronel 300 mg (Japan) | Placebo + Orteronel 200 mg (Ex-Japan) | Placebo + Orteronel 400 mg (Ex-Japan)
Started | 33 | 32 | 36 | 36
Completed | 0 | 0 | 0 | 0
Not Completed | 33 | 32 | 36 | 36
Not completed — Adverse Event | 3 | 13 | 7 | 7
Not completed — Progressive Disease | 11 | 9 | 19 | 20
Not completed — Symptomatic Deterioration | 1 | 0 | 2 | 0
Not completed — Unsatisfactory Therapeutic Response | 7 | 2 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 3
Not completed — Reason not Specified | 10 | 7 | 5 | 5

BASELINE CHARACTERISTICS:
Population: Data for baseline characteristics has been summarized as per the treatment received in Cycle 1.
Groups:
- Placebo + Orteronel 200 mg (Japan): Orteronel placebo-matching tablets, orally, twice daily (BID) in Cycle 1 (28 days) followed by orteronel 200 mg, tablets, orally, twice daily in 28 day cycles in Japan for up to 3 years. Study drug will be administered concomitantly with prednisone (or commercially available equivalent) 5 mg twice daily continuously throughout the study.
- Total: Total of all reporting groups
Arm/Group | Placebo + Orteronel 200 mg (Japan) | Orteronel 200 mg (Japan) | Placebo + Orteronel 300 mg (Japan) | Orteronel 300 mg (Japan) | Placebo + Orteronel 200 mg (Ex-Japan) | Orteronel 200 mg (Ex-Japan) | Placebo + Orteronel 400 mg (Ex-Japan) | Orteronel 400 mg (Ex-Japan) | Total
Number analyzed (Participants) | 11 | 22 | 10 | 22 | 11 | 25 | 12 | 24 | 137
Age, Continuous [Mean (Full Range); unit: years] | 72.1 [62 to 84] | 68.5 [52 to 82] | 70.1 [59 to 76] | 71.5 [51 to 85] | 69.6 [51 to 85] | 69.9 [55 to 84] | 73.3 [60 to 84] | 69.4 [49 to 88] | 70.6 [49 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 11 | 22 | 10 | 22 | 11 | 25 | 12 | 24 | 137
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 11 | 22 | 10 | 22 | 11 | 25 | 12 | 23 | 136
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 0 | 0 | 0 | 0 | 11 | 25 | 11 | 23 | 70
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Asian - Japanese | 11 | 22 | 10 | 22 | 0 | 0 | 0 | 0 | 65
Region of Enrollment [Number; unit: participants]
  Japan | 11 | 22 | 10 | 22 | 0 | 0 | 0 | 0 | 65
  Australia | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 2 | 8
  Greece | 0 | 0 | 0 | 0 | 2 | 4 | 1 | 3 | 10
  Ireland | 0 | 0 | 0 | 0 | 2 | 5 | 3 | 3 | 13
  Netherlands | 0 | 0 | 0 | 0 | 1 | 6 | 1 | 5 | 13
  United Kingdom | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3
  United States | 0 | 0 | 0 | 0 | 2 | 9 | 4 | 10 | 25
Height [Mean (Full Range); unit: cm] | 161.94 [153.0 to 168.2] | 167.10 [154.0 to 177.5] | 163.92 [156.6 to 170.7] | 164.71 [151.0 to 174.0] | 170.41 [157.0 to 184.7] | 174.79 [162.0 to 186.0] | 176.70 [165.0 to 185.4] | 174.74 [162.0 to 189.0] | 169.29 [151.0 to 189.0]
Weight [Mean (Full Range); unit: kg] | 65.82 [55.1 to 82.4] | 70.32 [47.5 to 85.2] | 65.75 [55.5 to 76.0] | 64.49 [44.7 to 87.1] | 87.34 [67.0 to 113.0] | 90.39 [64.0 to 130.7] | 88.23 [64.9 to 114.1] | 89.85 [63.0 to 134.6] | 77.77 [44.7 to 134.6]
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 25.05 [20.6 to 30.4] | 25.21 [17.8 to 31.2] | 24.43 [21.1 to 28.7] | 23.73 [16.7 to 32.0] | 29.85 [23.8 to 37.8] | 29.61 [22.1 to 40.3] | 28.37 [18.9 to 39.9] | 29.40 [22.9 to 40.2] | 26.96 [16.7 to 40.3]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serum Testosterone Levels Reduced to ≤ 2 ng/dL After 4 Weeks of Treatment in Japan
Description: Serum Ultra-sensitive testosterone was measured by liquid chromatography at a central laboratory.
Time Frame: Baseline and Week 4
Population: Pharmacodynamics-evaluable population was defined as participants with a baseline and at least 1 post-baseline pharmacodynamics measurement.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo (Japan): Orteronel placebo-matching tablets, orally, twice daily in Cycle 1. Study drug will be administered concomitantly with prednisone (or commercially available equivalent) 5 mg twice daily (BID) continuously throughout the study.
Arm/Group | Placebo (Japan) | Orteronel 300 mg (Japan)
Number analyzed (Participants) | 21 | 22
percentage of participants | 86.0 [63.7 to 97.0] | 100.0 [84.6 to 100.0]
Statistical Analysis 1: Comparison: Placebo (Japan) vs Orteronel 300 mg (Japan); Test type: Superiority or Other; p = 0.1078, Fisher Exact

2. Secondary Outcome: Percentage of Participants With Serum Testosterone Levels Reduced to ≤ 2 ng/dL in Ex-Japan
Description: Serum Ultra-sensitive testosterone was measured by liquid chromatography at a central laboratory.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo (Ex-Japan): Orteronel placebo-matching tablets, orally, twice daily in Cycle 1. Study drug will be administered concomitantly with prednisone (or commercially available equivalent) 5 mg twice daily (BID) continuously throughout the study.
Arm/Group | Placebo (Ex-Japan) | Orteronel 400 mg (Ex-Japan)
Number analyzed (Participants) | 23 | 24
percentage of participants | 48.0 [26.8 to 69.4] | 79.0 [57.8 to 92.9]
Statistical Analysis 1: Comparison: Placebo (Ex-Japan) vs Orteronel 400 mg (Ex-Japan); Test type: Superiority or Other; p = 0.0355, Fisher Exact; Odds Ratio (OR) = 4.145, 95% CI 2-sided [0.9895 to 18.7606] — Odds ratio >1 favors orteronel

3. Secondary Outcome: Percent Change From Baseline in Serum Testosterone Level After 4 Weeks of Treatment
Description: Serum Ultra-sensitive testosterone was measured by liquid chromatography at a central laboratory.
Time Frame: Baseline and Week 4
Population: Participants from the Pharmacodynamics-evaluable population, defined as participants with a baseline and at least 1 post-baseline pharmacodynamics measurement, with data available after 4 Weeks of Treatment.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Placebo (Japan): Orteronel placebo-matching tablets, orally, twice daily in Cycle 1 (28 days). Study drug will be administered concomitantly with prednisone (or commercially available equivalent) 5 mg twice daily (BID) continuously throughout the study.
Arm/Group | Placebo (Japan) | Orteronel 200 mg (Japan) | Orteronel 300 mg (Japan) | Placebo (Ex-Japan) | Orteronel 200 mg (Ex-Japan) | Orteronel 400 mg (Ex-Japan)
Number analyzed (Participants) | 21 | 22 | 22 | 20 | 21 | 22
percent change | -87.666 (10.4250) | -97.245 (1.2548) | -96.812 (2.7055) | -63.702 (43.3941) | -86.268 (37.2015) | -53.954 (118.8050)

4. Secondary Outcome: Percent Change From Baseline in Serum Testosterone Level After 12 Weeks of Treatment
Description: Serum Ultra-sensitive testosterone was measured by liquid chromatography at a central laboratory.
Time Frame: Baseline and Week 12
Population: Participants from the Pharmacodynamics-evaluable population, defined as participants with a baseline and at least 1 post-baseline pharmacodynamics measurement, with data available after 12 Weeks of Treatment.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Orteronel 200 mg (Japan) | Orteronel 300 mg (Japan) | Orteronel 200 mg (Ex-Japan) | Orteronel 400 mg (Ex-Japan)
Number analyzed (Participants) | 31 | 26 | 28 | 31
percent change | -95.804 (5.3367) | -95.703 (5.7468) | -91.311 (17.5217) | -14.442 (406.3116)

5. Secondary Outcome: Percentage of Participants With Prostate-Specific Antigen Reduction ≥ 50% (PSA50) After 4 Weeks of Treatment
Description: A 50% PSA response rate (PSA50) was defined as PSA reduction ≥ 50% from Baseline.
Time Frame: Baseline and Week 4
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Japan) | Orteronel 200 mg (Japan) | Orteronel 300 mg (Japan) | Placebo (Ex-Japan) | Orteronel 200 mg (Ex-Japan) | Orteronel 400 mg (Ex-Japan)
Number analyzed (Participants) | 21 | 22 | 22 | 23 | 25 | 24
percentage of participants | 48.0 [25.7 to 70.2] | 50.0 [28.2 to 71.8] | 41.0 [20.7 to 63.6] | 17.0 [5.0 to 38.8] | 48.0 [27.8 to 68.7] | 46.0 [25.6 to 67.2]

6. Secondary Outcome: Percentage of Participants With PSA50 After 12 Weeks of Treatment
Description: A 50% PSA response rate (PSA50) was defined as PSA reduction ≥ 50% from Baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Orteronel 200 mg (Japan) | Orteronel 300 mg (Japan) | Orteronel 200 mg (Ex-Japan) | Orteronel 400 mg (Ex-Japan)
Number analyzed (Participants) | 33 | 32 | 36 | 36
percentage of participants | 55.0 [36.4 to 71.9] | 47.0 [29.1 to 65.3] | 56.0 [38.1 to 72.1] | 44.0 [27.9 to 61.9]

7. Secondary Outcome: Absolute Values for Testosterone
Description: Serum Ultra-sensitive testosterone was measured by liquid chromatography at a central laboratory.
Time Frame: Baseline, Cycle 1 Day 8 and Cycle 2 Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Placebo (Japan) | Orteronel 200 mg (Japan) | Orteronel 300 mg (Japan) | Placebo (Ex-Japan) | Orteronel 200 mg (Ex-Japan) | Orteronel 400 mg (Ex-Japan)
Number analyzed (Participants) | 21 | 22 | 22 | 23 | 25 | 24
ng/dL
  Baseline | 9.749 (3.8460) | 9.079 (4.4581) | 10.148 (4.6504) | 9.173 (5.6123) | 9.263 (5.6572) | 14.588 (13.9833)
  Cycle 1 Day 8: number analyzed (Participants) | 20 | 22 | 22 | 19 | 20 | 21
  Cycle 1 Day 8 | 1.957 (2.2843) | 0.213 (0.0449) | 0.251 (0.1727) | 3.509 (4.3471) | 0.345 (0.2770) | 6.658 (20.4347)
  Cycle 2 Day 1: number analyzed (Participants) | 21 | 22 | 22 | 20 | 21 | 22
  Cycle 2 Day 1 | 1.096 (0.7751) | 0.203 (0.0145) | 0.270 (0.2311) | 3.095 (3.7254) | 0.266 (0.1837) | 11.720 (45.1753)

8. Secondary Outcome: Absolute Values for Dehydroepiandrosterone Sulfate (DHEA-S)
Description: Serum Ultra low level quantification of DHEA-S was measured by liquid chromatography and mass spectrometry (LC/MS) at a central laboratory.
Time Frame: Baseline, Cycle 1 Day 8 and Cycle 2 Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Placebo (Japan) | Orteronel 200 mg (Japan) | Orteronel 300 mg (Japan) | Placebo (Ex-Japan) | Orteronel 200 mg (Ex-Japan) | Orteronel 400 mg (Ex-Japan)
Number analyzed (Participants) | 21 | 22 | 22 | 23 | 25 | 24
nmol/L
  Baseline | 1928.0 (1306.59) | 2529.0 (1309.39) | 2340.9 (1606.36) | 2601.7 (3009.41) | 1783.0 (1554.76) | 2155.7 (1591.51)
  Cycle 1 Day 8: number analyzed (Participants) | 21 | 22 | 22 | 20 | 23 | 22
  Cycle 1 Day 8 | 414.9 (392.63) | 63.4 (55.11) | 71.8 (80.23) | 973.8 (1677.95) | 116.9 (161.01) | 226.6 (328.70)
  Cycle 2 Day 1: number analyzed (Participants) | 21 | 22 | 22 | 20 | 22 | 22
  Cycle 2 Day 1 | 268.9 (357.32) | 14.5 (21.83) | 36.3 (123.48) | 815.7 (1918.88) | 21.5 (25.68) | 180.6 (527.03)

9. Secondary Outcome: Absolute Values for Adrenocorticotropic Hormone (ACTH)
Description: Serum ACTH was measured by immunometric assay at the central laboratory.
Time Frame: Baseline, Cycle 1 Day 8 and Cycle 2 Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Placebo (Japan) | Orteronel 200 mg (Japan) | Orteronel 300 mg (Japan) | Placebo (Ex-Japan) | Orteronel 200 mg (Ex-Japan) | Orteronel 400 mg (Ex-Japan)
Number analyzed (Participants) | 21 | 22 | 22 | 23 | 25 | 24
pmol/L
  Baseline | 5.0 (1.66) | 5.5 (2.54) | 8.3 (4.98) | 4.7 (2.06) | 6.0 (4.05) | 6.4 (4.04)
  Cycle 1 Day 8: number analyzed (Participants) | 21 | 22 | 22 | 22 | 21 | 18
  Cycle 1 Day 8 | 3.1 (2.68) | 2.3 (1.55) | 3.0 (2.70) | 3.1 (2.62) | 3.8 (3.04) | 3.2 (2.56)
  Cycle 2 Day 1: number analyzed (Participants) | 21 | 22 | 22 | 22 | 24 | 22
  Cycle 2 Day 1 | 1.7 (1.19) | 1.7 (1.08) | 2.7 (2.17) | 3.0 (1.73) | 3.7 (4.38) | 3.6 (2.26)

10. Secondary Outcome: Absolute Values for Corticosterone
Description: Serum Corticosterone was measured by high pressure liquid chromatography with mass spectrometry at the central laboratory.
Time Frame: Baseline, Cycle 1 Day 8 and Cycle 2 Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Placebo (Japan) | Orteronel 200 mg (Japan) | Orteronel 300 mg (Japan) | Placebo (Ex-Japan) | Orteronel 200 mg (Ex-Japan) | Orteronel 400 mg (Ex-Japan)
Number analyzed (Participants) | 21 | 22 | 22 | 23 | 25 | 24
nmol/L
  Baseline | 5.946 (3.4433) | 6.515 (4.8246) | 7.768 (6.8625) | 6.317 (4.1467) | 10.030 (7.7341) | 17.975 (35.0695)
  Cycle 1 Day 8: number analyzed (Participants) | 21 | 22 | 22 | 20 | 23 | 21
  Cycle 1 Day 8 | 1.530 (1.6404) | 11.067 (14.4220) | 9.709 (13.4538) | 5.598 (7.1366) | 48.668 (66.3904) | 60.301 (77.5434)
  Cycle 2 Day 1: number analyzed (Participants) | 21 | 22 | 22 | 20 | 23 | 22
  Cycle 2 Day 1 | 0.758 (0.5108) | 11.108 (9.0708) | 14.654 (9.2064) | 4.321 (6.4063) | 29.929 (35.5565) | 47.204 (53.4566)

11. Secondary Outcome: Absolute Values for Cortisol
Description: Serum Cortisol was measured by immunometric assay at the central laboratory.
Time Frame: Baseline, Cycle 1 Day 8 and Cycle 2 Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Placebo (Japan) | Orteronel 200 mg (Japan) | Orteronel 300 mg (Japan) | Placebo (Ex-Japan) | Orteronel 200 mg (Ex-Japan) | Orteronel 400 mg (Ex-Japan)
Number analyzed (Participants) | 21 | 22 | 22 | 23 | 25 | 24
nmol/L
  Baseline | 366.5 (116.69) | 371.3 (119.38) | 383.4 (125.98) | 384.8 (117.14) | 449.0 (131.54) | 446.8 (193.09)
  Cycle 1 Day 8: number analyzed (Participants) | 21 | 22 | 22 | 23 | 24 | 22
  Cycle 1 Day 8 | 82.3 (46.16) | 49.5 (25.53) | 55.5 (55.97) | 175.8 (107.82) | 100.9 (87.38) | 122.0 (88.70)
  Cycle 2 Day 1: number analyzed (Participants) | 20 | 22 | 22 | 21 | 24 | 23
  Cycle 2 Day 1 | 53.9 (24.92) | 49.2 (21.71) | 54.3 (39.93) | 149.6 (122.91) | 97.2 (85.66) | 109.1 (83.19)

12. Secondary Outcome: Absolute Values for Prostate-Specific Antigen (PSA)
Description: Serum PSA was measured at the central laboratory.
Time Frame: Baseline and Cycle 2 Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo (Japan) | Orteronel 200 mg (Japan) | Orteronel 300 mg (Japan) | Placebo (Ex-Japan) | Orteronel 200 mg (Ex-Japan) | Orteronel 400 mg (Ex-Japan)
Number analyzed (Participants) | 21 | 22 | 22 | 23 | 25 | 24
ng/mL
  Baseline | 37.588 (48.9413) | 27.227 (24.8821) | 97.504 (293.9496) | 133.238 (189.9345) | 165.992 (368.5016) | 100.237 (210.5675)
  Cycle 2 Day 1: number analyzed (Participants) | 20 | 22 | 22 | 21 | 24 | 23
  Cycle 2 Day 1 | 24.325 (46.9725) | 18.005 (16.9858) | 38.892 (95.0124) | 152.940 (261.9735) | 117.257 (286.1870) | 56.437 (97.1621)

13. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Orteronel and M-I Metabolite
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: Cycle 1 Day 1 Predose, 0.5, 1, 2, 3, 5, 8, 12 hours post-dose
Population: Pharmacokinetic Population included all randomized participants who received orteronel in Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Orteronel 200 mg (Japan) | Orteronel 300 mg (Japan) | Orteronel 200 mg (Ex-Japan) | Orteronel 400 mg (Ex-Japan)
Number analyzed (Participants) | 22 | 22 | 25 | 24
ng/mL
  Orteronel | 1520 (23.9) | 2210 (33.9) | 1300 (59.7) | 1610 (50.3)
  Orteronel Metabolite M-I | 272 (33.1) | 422 (37.0) | 199 (61.9) | 261 (47.2)

14. Secondary Outcome: AUC(0-12): Area Under the Plasma Concentration-Time Curve From Time 0 to 12 Hours Post-dose for Orteronel and M-I Metabolite
Description: AUC(0-12) is measure of area under the curve over the dosing interval where the length of the dosing interval is time 0 to 12 hours in this study.
Time Frame: Cycle 1 Day 1 Predose, 0.5, 1, 2, 3, 5, 8, 12 hours post-dose
Population: Pharmacokinetic Population included all randomized participants who received orteronel in Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Orteronel 200 mg (Japan) | Orteronel 300 mg (Japan) | Orteronel 200 mg (Ex-Japan) | Orteronel 400 mg (Ex-Japan)
Number analyzed (Participants) | 22 | 22 | 25 | 24
h*ng/mL
  Orteronel | 8810 (16.4) | 12800 (31.2) | 7830 (51.1) | 10200 (41.4)
  Orteronel Metabolite M-I | 2130 (28.3) | 3290 (33.8) | 1570 (65.5) | 2080 (44.8)

15. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Orteronel and M-I Metabolite
Description: Tmax: Time to reach the maximum plasma concentration (Cmax), equal to time (hours) to Cmax.
Time Frame: Cycle 1 Day 1 Predose, 0.5, 1, 2, 3, 5, 8, 12 hours post-dose
Population: Pharmacokinetic Population included all randomized participants who received orteronel in Cycle 1.
Measure: Median (Full Range); unit: hours
Arm/Group | Orteronel 200 mg (Japan) | Orteronel 300 mg (Japan) | Orteronel 200 mg (Ex-Japan) | Orteronel 400 mg (Ex-Japan)
Number analyzed (Participants) | 22 | 22 | 25 | 24
hours
  Orteronel | 2.97 [1.00 to 5.10] | 2.43 [1.00 to 4.97] | 2.00 [0.500 to 7.93] | 1.92 [0.500 to 5.00]
  Orteronel Metabolite M-I | 5.00 [2.03 to 8.10] | 4.98 [2.00 to 8.23] | 5.05 [1.03 to 11.1] | 4.98 [1.22 to 11.2]

16. Secondary Outcome: AE (0-24) Cumulative Amount of Drug Excreted Into the Urine for Orteronel and MI-Metabolite
Description: Cumulative amount of urine excreted time 0 to 24 hour.
Time Frame: Cycle 1 Day 1 Predose, 0.5, 1, 2, 3, 5, 8, 12 hours post-dose
Population: Pharmacokinetic Population included all randomized participants who received orteronel in Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Orteronel 200 mg (Japan) | Orteronel 300 mg (Japan) | Orteronel 200 mg (Ex-Japan) | Orteronel 400 mg (Ex-Japan)
Number analyzed (Participants) | 22 | 22 | 25 | 24
mg
  Orteronel | 115.0 (26.0) | 164.0 (26.2) | 95.3 (31.9) | 161.0 (41.4)
  Orteronel Metabolite M-I | 39.6 (31.5) | 62.5 (26.6) | 30.0 (40.1) | 52.8 (46.4)

17. Secondary Outcome: Cmax,ss: Maximum Observed Plasma Concentration at Steady State for Orteronel and MI-Metabolite
Description: Maximum observed steady-state plasma concentration during a dosing interval.
Time Frame: Cycle 1 Day 8 Predose, 0.5, 1, 2, 3, 5, 8, 12 hours post-dose
Population: Pharmacokinetic Population included all randomized participants who received orteronel in Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Orteronel 200 mg (Japan) | Orteronel 300 mg (Japan) | Orteronel 200 mg (Ex-Japan) | Orteronel 400 mg (Ex-Japan)
Number analyzed (Participants) | 22 | 22 | 25 | 24
ng/mL
  Orteronel | 2180 (22.4) | 3210 (31.5) | 1840 (37.1) | 3100 (45.0)
  Orteronel Metabolite M-I | 565 (32.4) | 864 (39.5) | 485 (75.4) | 761 (81.3)

18. Secondary Outcome: Tmax,ss: Time to Reach the Maximum Plasma Concentration (Cmax), Equal to Time (Hours) to Cmax at Steady State for Orteronel and M-I Metabolite
Description: Time to reach the maximum plasma concentration (Cmax), equal to time (hours) to Cmax at steady state.
Time Frame: Cycle 1 Day 8 Predose, 0.5, 1, 2, 3, 5, 8, 12 hours post-dose
Population: Pharmacokinetic Population included all randomized participants who received orteronel in Cycle 1.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Orteronel 200 mg (Japan) | Orteronel 300 mg (Japan) | Orteronel 200 mg (Ex-Japan) | Orteronel 400 mg (Ex-Japan)
Number analyzed (Participants) | 22 | 22 | 25 | 24
hours
  Orteronel | 2.05 [1.00 to 5.08] | 2.96 [1.00 to 5.17] | 2.00 [0.550 to 5.17] | 1.98 [0.500 to 3.08]
  Orteronel Metabolite M-I | 3.08 [2.00 to 5.17] | 4.78 [2.00 to 8.13] | 3.00 [1.00 to 5.07] | 3.00 [0 to 8.00]

19. Secondary Outcome: AUC(0-tau): Area Under the Plasma Concentration-time Curve From Time 0 to Time Tau Over the Dosing Interval for Orteronel and M-I Metabolite
Description: Area under the plasma concentration-time curve during a dosing interval, where tau is the length of the dosing interval.
Time Frame: Cycle 1 Day 8 Predose, 0.5, 1, 2, 3, 5, 8, 12 hours post-dose
Population: Pharmacokinetic Population included all randomized participants who received orteronel in Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Orteronel 200 mg (Japan) | Orteronel 300 mg (Japan) | Orteronel 200 mg (Ex-Japan) | Orteronel 400 mg (Ex-Japan)
Number analyzed (Participants) | 22 | 22 | 25 | 24
h*ng/mL
  Orteronel | 13300 (20.4) | 20400 (36.1) | 12600 (36.2) | 20000 (55.0)
  Orteronel Metabolite M-I | 4840 (35.0) | 7460 (46.3) | 4340 (69.4) | 6590 (78.0)

20. Secondary Outcome: Rac: Accumulation Index for Orteronel and M-I Metabolite
Description: Rac was calculated as the ratio of AUCtau to AUC12hr.
Time Frame: Cycle 1 Day 8 Predose, 0.5, 1, 2, 3, 5, 8, 12 hours post-dose
Population: Pharmacokinetic Population included all randomized participants who received orteronel in Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Orteronel 200 mg (Japan) | Orteronel 300 mg (Japan) | Orteronel 200 mg (Ex-Japan) | Orteronel 400 mg (Ex-Japan)
Number analyzed (Participants) | 22 | 22 | 25 | 24
ratio
  Orteronel | 1.51 (9.1) | 1.59 (46.6) | 1.62 (39.3) | 1.97 (90.5)
  Orteronel Metabolite M-I | 2.27 (17.5) | 2.26 (43.0) | 2.76 (45.0) | 3.17 (77.7)

21. Secondary Outcome: Ctrough,ss: Observed Predose Plasma Concentration at Steady State for Orteronel and M-I Metabolite
Description: Observed predose plasma concentration at steady state.
Time Frame: Cycle 1 Day 8 Predose
Population: Pharmacokinetic Population included all randomized participants who received orteronel in Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Orteronel 200 mg (Japan) | Orteronel 300 mg (Japan) | Orteronel 200 mg (Ex-Japan) | Orteronel 400 mg (Ex-Japan)
Number analyzed (Participants) | 22 | 22 | 24 | 22
ng/mL
  Orteronel | 710 (28.1) | 1060 (63.7) | 807 (45.4) | 899 (59.8)
  Orteronel Metbolite M-I | 291 (47.1) | 444 (66.7) | 314 (68.6) | 417 (58.0)

22. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding),symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study A serious adverse event is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: From signing of the informed consent form through 30 days after the last dose of study drug, approximately 3.2 years
Population: Safety Population included all randomized participants who received at least one dose of study drug. Adverse events are summarized as per the treatment received.
Measure: Number; unit: participants
Groups:
- Orteronel 200 mg (Japan): Orteronel 200 mg, tablets, orally, twice daily in 28 day cycles in Japan and ex-Japan for up to 3 years. Study drug will be administered concomitantly with prednisone (or commercially available equivalent) 5 mg twice daily (BID) continuously throughout the study.
Arm/Group | Placebo (Japan) | Orteronel 200 mg (Japan) | Orteronel 300 mg (Japan) | Placebo (Ex-Japan) | Orteronel 200 mg (Ex-Japan) | Orteronel 400 mg (Ex-Japan)
Number analyzed (Participants) | 21 | 33 | 32 | 23 | 36 | 36
participants
  AE | 7 | 33 | 32 | 18 | 36 | 36
  SAE | 0 | 8 | 18 | 1 | 16 | 12

ADVERSE EVENTS:
Time Frame: From signing of the informed consent form through 30 days after the last dose of study drug, approximately 3.2 years.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Adverse events were summarized as per the treatment received.
Groups:
- Placebo: Orteronel placebo-matching tablets, orally, twice daily in Cycle 1 (28 days). Study drug will be administered concomitantly with prednisone (or commercially available equivalent) 5 mg twice daily (BID) continuously throughout the study.
- Orteronel 200 mg (Japan): Orteronel 200 mg, tablets, orally, twice daily in 28 day cycles in for up to 2.8 years. Study drug will be administered concomitantly with prednisone (or commercially available equivalent) 5 mg twice daily (BID) continuously throughout the study.
- Orteronel 200 mg (Ex-Japan): Orteronel 200 mg, tablets, orally, twice daily in 28 day cycles in for up to 3.1 years. Study drug will be administered concomitantly with prednisone (or commercially available equivalent) 5 mg twice daily (BID) continuously throughout the study.
- Orteronel 400mg (Ex-Japan): Orteronel 400 mg, tablets, orally, twice daily in 28 day cycles Ex-Japan for up to 3.1 years. Study drug will be administered concomitantly with prednisone (or commercially available equivalent) 5 mg twice daily (BID) continuously throughout the study.
Arm/Group | Placebo | Orteronel 200 mg (Japan) | Orteronel 300 mg (Japan) | Orteronel 200 mg (Ex-Japan) | Orteronel 400mg (Ex-Japan)
Serious Adverse Events (participants affected / at risk) | 10/44 | 8/33 | 18/32 | 16/36 | 12/36
Other Adverse Events (participants affected / at risk) | 44/44 | 33/33 | 32/32 | 35/36 | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=44) | Orteronel 200 mg (Japan) (N=33) | Orteronel 300 mg (Japan) (N=32) | Orteronel 200 mg (Ex-Japan) (N=36) | Orteronel 400mg (Ex-Japan) (N=36)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 2 (3) | 2 (2) | 2 (2)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pancreatic enzymes increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device occlusion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large Intestine Polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomitting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary Artery Stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial Ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile Duct Stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal Ligament Ossification (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Altered State Of Consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device Related Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Angiodysplasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal Colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Metastatic Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=44) | Orteronel 200 mg (Japan) (N=33) | Orteronel 300 mg (Japan) (N=32) | Orteronel 200 mg (Ex-Japan) (N=36) | Orteronel 400mg (Ex-Japan) (N=36)
Lipase increased (Investigations) | 19 (36) | 25 (46) | 19 (32) | 9 (10) | 7 (9)
Amylase increased (Investigations) | 16 (21) | 21 (35) | 19 (27) | 4 (7) | 6 (10)
Constipation (Gastrointestinal disorders) | 7 (7) | 8 (9) | 10 (12) | 10 (13) | 12 (13)
Diarrhoea (Gastrointestinal disorders) | 11 (12) | 4 (4) | 5 (6) | 15 (30) | 13 (16)
Fatigue (General disorders) | 8 (9) | 0 (0) | 2 (3) | 19 (22) | 15 (17)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 (16) | 3 (3) | 8 (9) | 8 (11) | 12 (22)
Nausea (Gastrointestinal disorders) | 7 (12) | 5 (6) | 7 (10) | 13 (17) | 12 (16)
Hot flush (Vascular disorders) | 7 (7) | 3 (3) | 5 (5) | 5 (5) | 10 (10)
Diabetes mellitus (Metabolism and nutrition disorders) | 5 (5) | 9 (10) | 6 (8) | 1 (1) | 4 (4)
Alanine aminotransferase increased (Investigations) | 6 (7) | 7 (7) | 7 (11) | 2 (4) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 6 (8) | 7 (7) | 7 (11) | 2 (4) | 1 (1)
Oedema peripheral (General disorders) | 4 (4) | 8 (10) | 6 (7) | 7 (7) | 5 (6)
Decreased appetite (Metabolism and nutrition disorders) | 5 (7) | 1 (1) | 5 (8) | 9 (10) | 7 (8)
Gamma-glutamyltransferase increased (Investigations) | 6 (6) | 5 (6) | 8 (14) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (4) | 3 (11) | 9 (12) | 3 (3)
Weight decreased (Investigations) | 5 (5) | 2 (2) | 6 (9) | 2 (2) | 3 (4)
Dysgeusia (Nervous system disorders) | 3 (3) | 2 (2) | 4 (4) | 4 (4) | 4 (4)
Hypertension (Vascular disorders) | 4 (4) | 3 (3) | 3 (3) | 2 (2) | 8 (8)
Nasopharyngitis (Infections and infestations) | 7 (7) | 8 (10) | 8 (13) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 5 (5) | 8 (8) | 4 (4) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2) | 2 (2) | 6 (6) | 4 (4)
Upper respiratory trat infection (Infections and infestations) | 4 (4) | 3 (4) | 4 (5) | 6 (7) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 4 (5) | 3 (3) | 5 (5)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4) | 4 (4) | 2 (3) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 3 (3) | 5 (6) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 2 (3) | 2 (2) | 1 (1) | 4 (4)
Malaise (General disorders) | 4 (5) | 4 (5) | 6 (7) | 3 (3) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0) | 5 (5) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 4 (5)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 3 (4) | 5 (8) | 2 (4) | 5 (6)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 4 (4) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 5 (6) | 4 (5)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 6 (7) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 1 (2) | 0 (0) | 4 (8) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 5 (5) | 4 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 2 (2) | 1 (3) | 2 (2)
Rash macular (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (4) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 0 (0) | 2 (2) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 2 (2) | 2 (2) | 3 (4) | 2 (7)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (4) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 3 (4) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 5 (6) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 4 (4) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (4) | 3 (4)
Nocturia (Renal and urinary disorders) | 3 (4) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (4) | 2 (4) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (4) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 3 (5) | 3 (4) | 3 (5) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (5)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Chronic Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Face Oedema (General disorders) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (3) | 1 (5) | 2 (3)
Cystitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3) | 3 (8) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (4) | 1 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (3)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.